CLINICAL TRIAL: NCT04328597
Title: Portuguese Inguinal Hernia Cohort Study
Brief Title: Portuguese Inguinal Hernia Cohort (PINE) Study
Acronym: PINE
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Portuguese Surgical Research Collaborative (Network)
Collaborators: University of Lisbon (Other)
Responsible Party: Sponsor
Other Study IDs: Version 1
Record Dates: First submitted 2020-03-25; First posted 2020-03-31 (Actual); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Inguinal Hernia; Chronic Pain
MeSH Terms: conditions — Hernia, Inguinal; Chronic Pain | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic postoperative pain: Patients scoring 3 or more on the EuraHS Quality of Life assessment after elective inguinal hernia repair
  Interventions: Procedure: Inguinal hernia repair
- Non chronic postoperative pain: Patients scoring less than 3 on the EuraHS Quality of Life assessment after elective inguinal hernia repair
  Interventions: Procedure: Inguinal hernia repair

INTERVENTIONS:
Procedure: Inguinal hernia repair — Inguinal hernia repair (open, laparo-endoscopic, robotic)
  Other Names: surgery

SUMMARY:
Prospective national cohort study of patients submitted to elective inguinal hernia repair. The primary outcome is the prevalence of chronic postoperative inguinal pain, according to the EuraHS QoL questionnaire at 3 months postoperatively. The study will be delivered in all Portuguese regions through a collaborative research network. Four 2-week inclusion periods will be open for recruitment. A site-specific questionnaire will capture procedure volume and logistical facilities for hernia surgery.

ELIGIBILITY:
Inclusion Criteria:

* Elective inguinal hernia repair in a portuguese hospital
* Willing and able to consent and comply with the follow up protocol

Exclusion Criteria:

* Urgent/emergent inguinal hernia repair

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Portuguese patients undergoing inguinal hernia repair in one of the hospitals participating in the study
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-10-07 (Actual); Primary Completion 2020-06-12 (Estimated); Study Completion 2020-08-12 (Estimated)

PRIMARY OUTCOMES:
Chronic postoperative pain | 3 months postoperatively
  Score of 3 or above on the pain domains of the European Registry for Abdominal Wall Hernias Quality of Life (EuraHS QoL) assessment, with higher scores indicating higher pain

SECONDARY OUTCOMES:
Proportion of patients receiving antibiotic prophylaxis before inguinal hernia repair | Intraoperatively
Proportion of patients operated as day case surgery | 30 days after surgery
Postoperative morbidity | 30 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Soares, Study Chair — Portuguese Surgical Research Collaborative
Locations (1):
- Hospital prof. Dr. Fernando Fonseca, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No
No plans are made to share patient data